CLINICAL TRIAL: NCT04719624
Title: Novel Porous Bioceramic Material as a Bone Substitute. Clinical Trial.
Brief Title: Novel Porous Bioceramic Material as a Bone Substitute
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Orton Orthopaedic Hospital (Other)
Collaborators: Biomendex Oy (Industry); Oral Hammaslääkärit Oy, Qmedical Pikku Huopalahti (Unknown); Tampere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AdaptosOral-001
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Alveolar Ridge Preservation
Keywords: synthetic bone graft; Adaptos; extraction socket; dental
MeSH Terms: interventions — Tooth Extraction; Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Adaptos-Si [0.5-1 mm] (Experimental): Bone augmentation, after tooth extraction, with Adaptos-Si [0.5-1 mm] (synthetic bone graft material) in combination with a gelatin sponge.
  Interventions: Device: Adaptos®-Si [0.5-1 mm] (bone grafting surgery)
- Adaptos-Si [1-2 mm] (Experimental): Bone augmentation, after tooth extraction, with Adaptos-Si [1-2 mm] (synthetic bone graft material) in combination with a gelatin sponge.
  Interventions: Device: Adaptos®-Si [1-2 mm] (bone grafting surgery)
- Bio-Oss (Active Comparator): Bone augmentation, after tooth extraction, with Bio-Oss (bovine-derived xenograft) in combination with a gelatin sponge.
  Interventions: Device: Geistlich Bio-Oss (bone grafting surgery)
- Empty extraction socket (Placebo Comparator): Post-extraction the socket filled only by clot.
  Interventions: Procedure: Tooth extraction without bone graft material
- Adaptos [1-2 mm] (Experimental): Bone augmentation, after tooth extraction, with Adaptos [1-2 mm] (synthetic bone graft material) in combination with a gelatin sponge.
  Interventions: Device: Adaptos® (bone grafting surgery)

INTERVENTIONS:
Device: Adaptos®-Si [0.5-1 mm] (bone grafting surgery) — After screening and enrollment, subjects will undergo tooth extraction of a single tooth with placement of one of the four randomized, synthetic bone graft substitutes with a gelatin sponge (Spongostan Dental). Following 5 months of healing a dental implant will be placed. The subjects will then be followed for another 5 months for healing. Follow-up visits will be at 2 weeks, 5 months, and 10 months.
  Other Names: Ridge preservation bone grafting after tooth extraction.
  Arms: Adaptos-Si [0.5-1 mm]
Device: Adaptos®-Si [1-2 mm] (bone grafting surgery) — After screening and enrollment, subjects will undergo tooth extraction of a single tooth with placement of one of the four randomized, synthetic bone graft substitutes with a gelatin sponge (Spongostan Dental). Following 5 months of healing a dental implant will be placed. The subjects will then be followed for another 5 months for healing. Follow-up visits will be at 2 weeks, 5 months, and 10 months.
  Other Names: Ridge preservation bone grafting after tooth extraction.
  Arms: Adaptos-Si [1-2 mm]
Device: Geistlich Bio-Oss (bone grafting surgery) — After screening and enrollment, subjects will undergo tooth extraction of a single tooth with placement of one of the four randomized, synthetic bone graft substitutes with a gelatin sponge (Spongostan Dental). Following 5 months of healing a dental implant will be placed. The subjects will then be followed for another 5 months for healing. Follow-up visits will be at 2 weeks, 5 months, and 10 months.
  Other Names: Ridge preservation bone grafting after tooth extraction.
  Arms: Bio-Oss
Procedure: Tooth extraction without bone graft material — After screening and enrollment, subjects will undergo tooth extraction of a single tooth and the socket is filled only by clot. Subject will be followed at 2 weeks, 5 months, and 10 months for healing.
  Arms: Empty extraction socket
Device: Adaptos® (bone grafting surgery) — After screening and enrollment, subjects will undergo tooth extraction of a single tooth with placement of one of the four randomized, synthetic bone graft substitutes with a gelatin sponge (Spongostan Dental). Following 5 months of healing a dental implant will be placed. The subjects will then be followed for another 5 months for healing. Follow-up visits will be at 2 weeks, 5 months, and 10 months.
  Other Names: Ridge preservation bone grafting after tooth extraction.
  Arms: Adaptos [1-2 mm]

SUMMARY:
The aim of this study is to demonstrate that new synthetic bone graft bioceramic composites (Adaptos®-Si and Adaptos®, Biomendex Oy) are able to support the preservation of the alveolar ridge and to promote bone regeneration following dental extraction. New bone graft substitutes are compared with already existing treatment principles used following dental extraction.

The primary hypothesis of the study is that Adaptos®-Si granules can reach a clinical outcome superior to that of dental socket left empty after extraction. Secondary aim is that new bioceramic composites can reach a clinical outcome non inferior to the active comparator of this study (Geistlisch Bio-Oss®).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate new synthetic Adaptos®-Si and Adaptos® in ridge preservation bone grafting after dental extraction. This is partly randomized, subject and outcome assessor-blinded, controlled, single center study. The total study duration for each patient is planned to be 10 months. In total 4 visits per patient are scheduled in this study.

Subjects will undergo a single tooth extraction and then will be randomized to receive one of the four bone graft substitutes, which are Adaptos®-Si (one of the the two granula sizes), Adaptos®, or Geistlich Bio-Oss®. Gelatin sponge is applied on the bone graft filled extraction socket. Non-randomized part of the study includes the patients that have chosen the conservative treatment option with dental socket left empty and no intention for dental implant placement. Following a healing period of 5 months, a dental implant will be placed, unless the patient has chosen the empty socket. The subject will be followed for ten months following tooth extraction. Bone ridge horizontal and vertical change assessment will be done by CBCT (primary and secondary outcome) at the time of tooth extraction, and 5 months and 10 months post-extraction.

The study device Bio-Oss® (Geistlich Pharma) and Spongostan Absorbable Haemostatic Gelatin Sponge (Ferrosan Medical Devices) are CE-marked. The products are used within the indication.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have voluntarily signed the informed consent
* Females and males, 18 years to 80 years of age
* Patient needs single tooth extraction of 1st or 2nd premolar or molar tooth
* At least one adjacent teeth present
* At least 3 intact walls
* Subjects must be committed to the study and the required follow-up visits

Exclusion Criteria:

* Planned radiation or radiation during previous year in the tooth extraction area.
* Smoking
* Osteoporosis
* Uncontrolled periodontitis
* Alcohol or drug abuse
* Pregnant or breastfeeding women
* Uncontrolled diabetes
* Local acute or chronic infection or presence of oral lesions or trauma
* Immunosuppressive disease, treatment, or medication
* Subject is part of the investigator team of this study or investigator's family member
* Subject is employee of one of the organizations involve in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge preservation, comparison between Adaptos-Si filled extraction sockets and empty sockets. | baseline, 5 months, and 10 months post-extraction
  Alveolar ridge horizontal and vertical change assessment by cone-beam computed tomography (CBCT). The vertical reference line is outlined from the apex through the center of the socket and the horizontal reference line through the apex perpendicular to the vertical line. The ridge width (in mm) is measured parallel to the horizontal reference line 1 mm, 3 mm, and 5 mm from the highest buccal ridge point on baseline. Ridge heights (in mm) are measured from the most apical point of the alveolar socket parallel to the vertical reference line. The dimensional changes of the ridge assessed on CBCT images immediately post-extraction, are acquired five months and ten months later. Comparison between Adaptos-Si filled extraction sockets and empty sockets.

SECONDARY OUTCOMES:
Alveolar ridge horizontal and vertical change (in mm) assessment by CBCT, comparisons between extraction sockets filled with Adaptos-Si or Bio-Oss bone graft substitutes. | baseline, 5 months, and 10 months post-extraction
  Alveolar ridge horizontal and vertical change assessment by cone-beam computed tomography (CBCT). The vertical reference line is outlined from the apex through the center of the socket and the horizontal reference line through the apex perpendicular to the vertical line. The ridge width (in mm) is measured parallel to the horizontal reference line 1 mm, 3 mm, and 5 mm from the highest buccal ridge point on baseline. Ridge heights (in mm) are measured from the most apical point of the alveolar socket parallel to the vertical reference line. The dimensional changes of the ridge assessed on CBCT images immediately post-extraction, are acquired five months and ten months later. Comparison between extraction sockets filled with Adaptos-Si or Bio-Oss bone graft substitutes.
Alveolar ridge horizontal and vertical change (in mm) assessment by CBCT, comparison between Adaptos filled extraction sockets and empty sockets. | baseline, 5 months, and 10 months post-extraction
  Alveolar ridge horizontal and vertical change assessment by cone-beam computed tomography (CBCT). The vertical reference line is outlined from the apex through the center of the socket and the horizontal reference line through the apex perpendicular to the vertical line. The ridge width (in mm) is measured parallel to the horizontal reference line 1 mm, 3 mm, and 5 mm from the highest buccal ridge point on baseline. Ridge heights (in mm) are measured from the most apical point of the alveolar socket parallel to the vertical reference line. The dimensional changes of the ridge assessed on CBCT images immediately post-extraction, are acquired five months and ten months later. Comparison between Adaptos filled extraction sockets and empty sockets.
Alveolar ridge horizontal and vertical change (in mm) assessment by CBCT, comparison between extraction sockets filled with Adaptos-Si or Adaptos bone graft substitutes. | baseline, 5 months, and 10 months post-extraction
  Alveolar ridge horizontal and vertical change assessment by cone-beam computed tomography (CBCT). The vertical reference line is outlined from the apex through the center of the socket and the horizontal reference line through the apex perpendicular to the vertical line. The ridge width (in mm) is measured parallel to the horizontal reference line 1 mm, 3 mm, and 5 mm from the highest buccal ridge point on baseline. Ridge heights (in mm) are measured from the most apical point of the alveolar socket parallel to the vertical reference line. The dimensional changes of the ridge assessed on CBCT images immediately post-extraction, are acquired five months and ten months later. Comparison between extraction sockets filled with Adaptos-Si or Adaptos bone graft substitutes.

OTHER OUTCOMES:
Comparison between radiological assessment methods | baseline, 5 months, and 10 months post-extraction
  The ridge width and height are measured from 2D images of CBCT scans (in mm) and change in dimensions in time is determined using these measurements. Reduction is also measured directly on the superimposed baseline and follow-up CBCT scans (in mm).The vertical reference line is outlined from the apex through the center of the socket and the horizontal reference line through the apex perpendicular to the vertical line. The ridge width (in mm) is measured parallel to the horizontal reference line 1 mm, 3 mm, and 5 mm from the highest buccal ridge point on baseline. Ridge heights (in mm) are measured from the most apical point of the alveolar socket parallel to the vertical reference line.

CONTACTS AND LOCATIONS:
Overall Officials: Antero Salo, MD, DDS, PhD, Principal Investigator — Oral Hammaslääkärit Oy, Qmedical Pikku Huopalahti
Locations (1):
- Oral Hammaslääkärit Oyj, Qmedical Pikku Huopalahti, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No